CLINICAL TRIAL: NCT05472922
Title: The Banded Mini Gastric Bypass Trial: A Prospective Randomized Controlled Trial
Acronym: RiMini
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marc van Det (Other)
Collaborators: Ziekenhuisgroep Twente (Other)
Responsible Party: Sponsor-Investigator, Marc van Det, principal investigator, Ziekenhuisgroep Twente
Organization: Ziekenhuisgroep Twente (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R22.025
Record Dates: First submitted 2022-06-22; First posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Bariatric Surgery; Weight Loss; Comorbidities and Coexisting Conditions
Keywords: MGB-OAGB; MiniMizer Ring; banded bypass
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Intervention Model Description: Non-blinded prospective randomized controlled single center trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Banded Mini Gastric Bypass (Experimental): Patients are treated for morbid obesity with a Mini gastric bypass (MGB-OAGB) with addition of the implantation of a MiniMizer Gastric Ring (Bariatric Solutions GmbH, Stein am Rhein Switzerland)
  Interventions: Device: Placement of MiniMizer Gastric Ring
- non-Banded Mini Gastric Bypass (Active Comparator): Patients are treated for morbid obesity with a Mini gastric bypass (MGB-OAGB)
  Interventions: Procedure: Normal MGB-OAGB

INTERVENTIONS:
Device: Placement of MiniMizer Gastric Ring — Insertion of MiniMizer Gastric Ring in addition to the normal MGB-OAGB
  Arms: Banded Mini Gastric Bypass
Procedure: Normal MGB-OAGB — No insertion of Minimizer Gastric Ring in addition to the normal MGB-OAGB
  Arms: non-Banded Mini Gastric Bypass

SUMMARY:
Rationale: Investigate if there is a significant weight reduction expressed in total body weight loss percentage (%TBWL) in patients 5 years after surgery, whom underwent a mini gastric bypass (MGB-OAGB) with addition of the implantation of a MiniMizer Ring.

Study design: A prospective non blinded single centre randomized controlled trial.

Sudy population: The study population will exist of patients eligible for MGB-OAGB surgery. Patients are invited to participate if Body Mass Index (BMI) ≥ 35kg/m2 with a comorbidity related to morbid obesity, or a BMI exceeding 40kg/m2.

Intervention: Insertion of the MiniMizer Ring around the gastric pouch in addition to the 'standard' MGB-OAGB.

Main study parameters/endpoints:

Primary Objective:

1. %TBWL 5 years after surgery.

   Secondary Objectives:
2. Percentage Excess Weight Loss (%EWL) 5 years after surgery.
3. Decrease or reduction of comorbidities (diabetes mellitus, hypertension, hyperlipidemia, sleep apnoea, and joint complaints).
4. Improvement of quality of life: SF-36 and OBESI-Q questionnaires.
5. Incidence and severity of dumping syndrome.
6. Incidence and severity of reflux symptoms: GERD-HRQoL questionnaire.
7. Incidence and complications due to silicone band.

Measurement of objectives are before surgery and six times after surgery combined with the standard postoperative care for patients who undergo bariatric surgery:

Expected advantages of bOLGB versus OLGB:

1. Increase of weight reduction, and due to that decrease of comorbidities and/or mortality related to overweight.
2. Long term decrease of weight regain.
3. Decrease of incidence of dumping.

Possible disadvantages of bOLGB versus OLGB:

1. Band-related complications such as erosion, infection, stenosis, or pouch dilatation.
2. Functional gastro-intestinal complains such as dysphagia and reflux.

ELIGIBILITY:
Inclusion Criteria:

* Patients meet IFSO criteria for Bariatric Surgery
* Age 18 and above

Exclusion Criteria:

* Previous Bariatric surgery
* Inability to read and understand written information
* Any genetic condition that can hamper the acceptance of medical advice
* chronic bowel disease
* Severe kidney of liver disease
* Pregnancy at the start or during the research period
* Patients with pre-existing therapy refractory GERD
* Patients with an allergy to silicone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Total Body Weight Change 5 years after surgery | 5 Years
  Percentage total body weight change 5 years after the procedure

SECONDARY OUTCOMES:
Change in Percentage Excess Weight (%EWL) 5 years after surgery | 5 years
  Change in Percentage Excess Weight (%EWL)
Change in (existing) co-morbidities 5 years after surgery | 5 years
  Change in severity of obesity-related co-morbidities: Type 2 Diabetes Mellitus (changes in HbA1c or use of antidiabetic medication), Hypertension (changes in bloodpressure or changes in use of antihypertensives), Osteo-arthritis (changes in VAS-score or use of analgesia drugs) , Hyperlipidemia (changes in HDL/LDL ratio, triglycerides or use of statine drugs), Obstructive Sleep Apnea syndrome (changes in use of CPEP treatment or changes is apneu hypopneu idex), and Gastro-Esophageal Reflux Disease (Changes in outcomes of GERD-HR questionnnaire which scoring scale runs from 0 (asymptomatic) to 50 (complete prohibitive) or changes in use of protonpompinhibitors)
Outcome measurement of SF-36 questionnaire | 5 years
  Evalution of changes in outcome of SF-36 Questionnaire 5 years after surgery. Scoring scale is described between 0 (lowest) and 100 (highest) to evaluate patient's welfare
Outcome measurement of OBESI-Q questionnaire | 5 years
  Evalution of changes in outcome of OBESI-Q Questionnaire 5 years after surgery. Scoring scale is described between 0 (lowest) and 100 (highest) to evaluate patient's welfare
Dumping Syndrome | 5 years
  The presence and severity of complains related to Dumping Syndrome in participants (yes or no)
Complications | 5 years
  The occurrence of short- and long-term complications of the minimizer ring

CONTACTS AND LOCATIONS:
Overall Officials: Marc J van Det, MD PhD, Principal Investigator — ZiekenhuisGroup Twente
Locations (1):
- Ziekenhuisgroep Twente, Almelo, Netherlands

IPD SHARING:
Plan to Share IPD: No
Individual Participant data will not be shared.

REFERENCES:
- [Derived] Tissink M, Verhagen T, Faneyte I, Hazebroek E, Oost S, Timmerman J, Veldhuis A, van Det M. The Banded One-Anastomosis Gastric Bypass Trial (RiMini Trial): Protocol of a Prospective Single-Center Randomized Controlled Trial. Obes Surg. 2025 May;35(5):1854-1859. doi: 10.1007/s11695-025-07751-6. Epub 2025 Mar 14. PMID 40085187